CLINICAL TRIAL: NCT00692289
Title: Quality of Life Analysis of Arimidex Treatment in Postmenopausal Patients With Breast Cancer
Acronym: RADAR II E
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OHU-ARI-2007/1
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an open label, non-interventional quality of life analysis for Arimidex treated postmenopausal patients in early breast cancer by investigator's questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Postmenopausal, hormon receptor positive patients with early breast cancer treated with Arimidex
* Investigators are requested to recruit patients only with at least 1 month prior Arimidex treatment.

Exclusion Criteria:

* Allergy to substance of medication
* Pre-perimenopausal woman
* Woman not eligible for treatment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal, hormonreceptor positive patients with early breast cancer treated with Arimidex (in accordance with the local SmPC).
Sampling Method: Non-Probability Sample
Enrollment: 1510 (Actual)
Dates: Start 2008-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Elements of the investigator questionnaire SF RAND-36 questionnaire | Quarterly (plus or minus 3 days )

SECONDARY OUTCOMES:
Investigator Assessment Report | Yearly (plus or minus 1 week )

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Horváth, M.D., Principal Investigator — National Institute of Oncology; Csaba Csongvai, Study Director — AstraZeneca Hungary; Éva Gulyás, Study Chair — AstraZeneca Hungary
Locations (6):
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Komló
  - Research Site, Miskolc
  - Research Site, Mohács
  - Research Site, Vác
  - Research Site, Zalaegerszeg